CLINICAL TRIAL: NCT04084847
Title: Effect of Berberis Vulgaris Consumption on Blood Pressure and Plasma Lipids in Subjects With Cardiovascular Risk Factors
Brief Title: Berberis Vulgaris Consumption and Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, Javad Nasrollahzadeh, Director, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 895
Record Dates: First submitted 2019-09-03; First posted 2019-09-10 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Blood Pressure; Cardiovascular Risk Factor; Lipid Profile
Keywords: Barberry; Berberis vulgaris; Blood pressure; Lipids; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Barberry (Active Comparator): Daily consumption of barberry in powder form.
  Interventions: Dietary Supplement: berberis vulgaris=barberry
- placebo (Placebo Comparator): Daily consumption of placebo powder.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: berberis vulgaris=barberry — 10 grams of barberry powder will be consumed daily for 8 weeks.
  Arms: Barberry
Dietary Supplement: Placebo — Placebo powder
  Arms: placebo

SUMMARY:
The aim of this study is to investigate the effect of barberry consumption on systolic and diastolic blood pressure, serum lipids, and inflammatory status. The study will involve cases having elevated BP (129/ < 85) and known hypertensive patients on medical treatment. Seventy people will be randomized into two groups, including intervention (barberry) or placebo groups.

Before and after of 8 week intervention, 24-hour ambulatory blood pressure monitoring will be done and fasting venous blood sample will be taken to measure plasma lipids. In addition, 24-hour urine will be collected to measure its sodium content and estimate sodium intake.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate in the study
* age between 20-65 years
* having elevated BP (129/ < 85) and known hypertensive patients on medical treatment
* at least one other classical cardiovascular disease risk factors, including hyperlipidemia or diabetes mellitus

Exclusion Criteria:

* Unwillingness to continue participation
* BMI> 30
* patients on nitrates
* high doses of statins consumption (Atorvastatin>40 mg/day or Rosuvastatin>20 mg/day)
* consumption of vitamins or minerals supplements during past month
* Chronic kidney disease stage 4 or 5

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
blood pressure | at 8 weeks
  mean of systolic and diastolic blood pressure of participants measured by ambulatory 24 hour blood pressure monitoring

SECONDARY OUTCOMES:
lipid profile | at 8 weeks
  plasma TC, LDL-C, HDL-C, TG
plasma NOx | at 8 weeks
  concentration of nitrite and nitrate in plasma
Inflammatory cytokine | at 8 weeks
  Plasma Interleukin-6

CONTACTS AND LOCATIONS:
Locations (1):
- Rajaei Cardiovascular, Medical & Research Center, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Emamat H, Zahedmehr A, Asadian S, Nasrollahzadeh J. The effect of barberry (Berberis integerrima) on lipid profile and systemic inflammation in subjects with cardiovascular risk factors: a randomized controlled trial. BMC Complement Med Ther. 2022 Mar 7;22(1):59. doi: 10.1186/s12906-022-03539-8. PMID 35255880
- [Derived] Emamat H, Zahedmehr A, Asadian S, Tangestani H, Nasrollahzadeh J. Effect of barberry (Berberis vulgaris) consumption on blood pressure, plasma lipids, and inflammation in patients with hypertension and other cardiovascular risk factors: study protocol for a randomized clinical trial. Trials. 2020 Nov 27;21(1):986. doi: 10.1186/s13063-020-04918-7. PMID 33246500